CLINICAL TRIAL: NCT04369521
Title: Evaluation of the Effects of a Low Free Sugar Diet on Lipid Profile, Glycemic Indices, Liver Enzymes, Inflammatory Factors and Hepatic Steatosis and Fibrosis in Patients With Nonalcoholic Fatty Liver Disease
Brief Title: Evaluation of the Effects of a Low Free Sugar Diet in Patients With Nonalcoholic Fatty Liver Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, Dr Azita Hekmatdoost, principal investigator, National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22300
Record Dates: First submitted 2020-04-27; First posted 2020-04-30 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Nonalcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): low free sugar diet with nutrition and exercise recommendation
  Interventions: Other: low free sugar diet
- control (No Intervention): regular diet with nutrition and exercise recommendation

INTERVENTIONS:
Other: low free sugar diet — low free sugar diet with nutrition and exercise recommendation
  Arms: Intervention

SUMMARY:
To study the effects of a low free sugar diet on lipid profile, glycemic indices, liver enzymes, inflammatory factors and hepatic steatosis and fibrosis in patients with Nonalcoholic fatty liver disease, 50 patients who referred to Gastrointestinal (GI) clinic with steatosis grade 2 and 3 will be randomly allocated to receive low free sugar diet or regular diet for 12 weeks; both groups will be advised to adherence the investigators' nutrition recommendation and exercise program too. At the first and the end of the intervention, lipid profiles, liver enzymes,glycemic indices, some inflammatory markers, and liver fibrosis will be assessed and compared between groups.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 to 60 years
2. Body Mass Index (BMI) between 25-40
3. Sonographic findings compatible with hepatic steatosis (degree 2 or more)

Exclusion Criteria:

1. Alcohol consumption
2. pregnancy or lactation
3. Other liver disease (viral,cirrhosis,...)
4. Use of drugs such as phenytoin,tamoxifen,lithium
5. A history of Cancer, autoimmune disease,Renal disease & Celiac disease, hypothyroidism or Cushing's syndrome
6. Lack of desire to continue studying
7. Have to use antibiotics with hepatotoxic drugs while studying
8. Non-compliance with diet

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-10-23 (Actual); Primary Completion 2020-05-09 (Estimated); Study Completion 2020-07-21 (Estimated)

PRIMARY OUTCOMES:
ALT | 12 weeks
  serum level of Alanine transaminase
AST | 12 weeks
  serum level of Aspartate transaminase
GGT | 12 weeks
  serum level of Gamma glutaminase
TG | 12 weeks
  serum level of Triglyceride
Total cholesterol | 12 weeks
  serum level of total cholesterol
LDL-c | 12 weeks
  serum level of LDL-Cholesterol
HDL-c | 12 weeks
  serum level of HDL-Cholesterol
FBS | 12 weeks
  serum level of Fasting blood sugar
Insulin | 12 weeks
  serum level of Insulin
hs-CRP | 12 weeks
  Serum level of high-sensitive C-reactive protein
TNF-a | 12 weeks
  Serum level of Tumor necrosis factor-a
NF-kb | 12 weeks
  Activity of Nuclear factor-B in peripheral monocellular cells
Liver fibrosis | 12 weeks
  Liver fibrosis according to fibroscan exam

CONTACTS AND LOCATIONS:
Locations (2):
- Iran (2):
  - Azita Hekmatdoost, Tehran, Middle East
  - National Nutrition and Food Technology Research Institute, Tehran